CLINICAL TRIAL: NCT03484065
Title: Quality of Life in Patients With Congenital Afibrinogenemia
Acronym: QualyAFIB
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Casini Alessandro, MD, University Hospital, Geneva
Other Study IDs: 2016-00447
Record Dates: First submitted 2018-03-14; First posted 2018-03-30 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Afibrinogenemia, Congenital
Keywords: Congenital fibrinogen disorders
MeSH Terms: conditions — Afibrinogenemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Afibrinogenemia
  Interventions: Other: Questionnaire quality of life

INTERVENTIONS:
Other: Questionnaire quality of life

SUMMARY:
The aim of this observational study is to evaluate the quality of life in patients with congenital afibrinogenemia using the Haemo-QoL SF for kids and the Haem-A-QoL for adult patients.

DETAILED DESCRIPTION:
In this observational study, children and adults suffering from congenital afibrinogenemia confirmed by biology will be enrolled. All patients will receive a questionnaire on quality of life in their own language during a routine visit and filled out by the patient at home. A general questionnaire will be filled out by the patient's physician.

ELIGIBILITY:
Inclusion Criteria:

* Congenital afibrinogenemia confirmed by biology (absence of circulating fibrinogen) and genotype

Exclusion Criteria:

* Lack of participant's consent
* Patient unable to understand the questionnaire

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients suffering from congenital afibrinogenemia
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
The influence of the afibrinogenemia on the patients' quality of life assessed by the Haemo-QoL SF questionnaire (for children) and the Haem-A-QoL questionnaire (for adult) | At inclusion
  The quality of life questionnaire includes item assessing:
  * Physical health
  * Feeling
  * View
  * Family
  * Friends
  * Others
  * Sport and school
  * Treatment
  * Perceived support
  * Dealing
  * Future
  * Relationship

SECONDARY OUTCOMES:
Impact of the afibrinogenemic patient's clinical phenotype on the patients' quality of life | At Inclusion
  The clinical phenotype will be assessed by a general questionnaire including data on:
  * Bleeding events
  * Bleeding events treatment
  * Thrombotic events
  * Thrombotic events treatment
  * Fibrinogen replacement (type of product and modality of replacement)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Casini, MD, Principal Investigator — University Hospitals of Geneva
Locations (28):
- United States (2):
  - Children's Hospital of Orange Count, Orange, California
  - Cohen Children's Medical Center, New Hyde Park, New York
- Béni Messous, Algiers, Algeria
- University of Calgary, Calgary, Canada
- Cairo University Pediatric Hospital, Cairo, Egypt
- Chru Lille, Lille, France
- Germany (2):
  - Universitats Kilinikum Frankfurt, Frankfurt
  - Dr von Haumer Children's Hospital, Munich
- India (2):
  - St John Medical College Hospital, Bangalore
  - All India Institute of Medical Sciences, New Delhi
- Sapienza Università di Roma, Roma, Italy
- University School of Medicine, Hamamatsu, Japan
- Kuwait University, Kuwait City, Kuwait
- Lebanon (2):
  - Hotel Dieu-de-France, Beirut
  - St George Hospital, Beirut
- Hopital d'Enfants de Rabat, Rabat, Morocco
- Radboud University Medical Centre, Nijmegen, Netherlands
- National Institute Of Blood Disease and Bone Marrow Transplantation, Karachi, Pakistan
- Institute of Hematology and Transfusion Medicine, Warsaw, Poland
- University Clinical Center, Belgrade, Serbia
- National Centre of Hemostasis and Thrombosis, Martin, Slovakia
- Hospital Universitari i Politecnic La Fe, Valencia, Spain
- Switzerland (2):
  - Inselspital, Bern
  - University Hospitals of Geneva, Geneva
- Hopital d'Enfants Bechir Hamza, Tunis, Tunisia
- Turkey (Türkiye) (3):
  - Uludag University, Bursa
  - Cerrahpasa Faculty of Medicine, Istanbul
  - Erciyes University, Kayseri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casini A, von Mackensen S, Santoro C, Djambas Khayat C, Belhani M, Ross C, Dorgalaleh A, Naz A, Unal E, Abdelwahab M, Lozeron ED, Trillot N, Susen S, Peyvandi F, de Moerloose P; QualyAfib Study Group. Clinical phenotype, fibrinogen supplementation, and health-related quality of life in patients with afibrinogenemia. Blood. 2021 Jun 3;137(22):3127-3136. doi: 10.1182/blood.2020009472. PMID 33512441